CLINICAL TRIAL: NCT01257880
Title: Comorbidities Associated With Migraine and Patent Foramen Ovale (CAMP)
Acronym: CAMP
Status: Completed | Type: Observational
Sponsor: Swedish Medical Center (Other)
Collaborators: University of Washington (Other); Coherex Medical (Industry); The John L. Locke, Jr. Charitable Trust (Unknown); National Headache Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 4865S-09
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Migraine With Aura; Patent Foramen Ovale
Keywords: Migraine; Migraine with Aura; Aura; Patent Foramen Ovale; Platelets; Sleep Apnea; Cognitive Function
MeSH Terms: conditions — Migraine with Aura; Foramen Ovale, Patent; Migraine Disorders; Epilepsy; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control (absence of PFO): Persons who have migraine aura and no evidence of PFO, based on transcranial Doppler evaluation.
- Large PFO: Persons who have migraine aura and large PFO, as assessed by transcranial Doppler evaluation.

SUMMARY:
The purpose of the study is to compare the rate of comorbidities associated with migraine aura (MA) between persons who have a large circulatory right-to-left shunt (RLS) and those who do not have RLS.

Approximately 50% of individuals who have MA also have RLS due to patent foramen ovale (PFO). A PFO is an anatomical opening or flap between the upper chambers of the heart or atria that permits blood to pass from the right of the heart to the left side of the heart, without first going to the lungs to be filtered and oxygenated. Many health conditions and clinical syndromes including stroke, sleep apnea, and migraine have been linked to PFO. Although the mechanism is undetermined, it is hypothesized that microscopic blood clots and chemicals such as serotonin can pass through the PFO, travel to the brain, and cause headache and aura.

Persons who have MA are at increased risk for stroke and transient ischemic attacks relative to people who do not have migraine. Migraine is also associated with the presence of white matter lesions in the brain and mild deficits in cognitive function associated with the posterior brain (vision, memory, processing speed). The risk of stroke in migraine is highest for women under the age of 45 who have aura and a high number of migraine headache days per month. No convincing evidence has been produced to explain the mechanism for the increased risk of ischemic stroke in migraine; however, increased platelet activation and aggregation is a plausible theory.

We hypothesize that migraineurs with aura and large RLS (presumably due to a PFO) will be more likely to have sleep apnea, increased platelet activation, cognitive deficits, alterations in cerebral vasomotor function, and white matter lesions than migraineurs with aura who do not have PFO. The results of this exploratory study will generate hypotheses as to why subgroups of migraineurs have an increased risk of stroke and the impact of large PFO on comorbid conditions associated with migraine aura. Early identification of migraine subgroups with a constellation of clinical syndromes that increase risk of neurovascular diseases will allow initiation of preventive strategies that may ultimately reduce burden and improve the productive quality of life for these individuals.

DETAILED DESCRIPTION:
A two-group observational study will be performed to determine if comorbidities associated with MA are more prevalent in the setting of large PFO. Potential subjects will be screened to assure that initial inclusion criteria are met (age, diagnosis of MA, monthly migraine frequency). Those who meet criteria will complete questionnaires including general medical history, migraine and aura frequencies, migraine-related disability, and treatment and preventive medications. In addition, subjects will be asked to complete two surveys on insomnia and sleep quality. Presence or absence of large PFO will be assessed by transcranial Doppler (TCD) bubble test. Subjects will also be screened for arterial variations in the Circle of Willis ("fetal origins") and carotid artery stenosis by duplex ultrasound examination of the arteries of the head and neck. If a subject is found to have a small-to-medium PFO on TCD evaluation, fetal origins, or carotid artery stenosis, s/he will be excluded from remaining study procedures.

Subjects who have either a large PFO or no PFO will undergo measurement of brain blood flow dynamics using TCD and carbon dioxide (CO2) stimulation to assess cerebral vasomotor reactivity. A blood specimen will be collected to assess three platelet activation biomarkers including CD40 ligand (sCD40L), P-selectin, and thromboxane B2 (TXB2). Subjects will be screened for sleep apnea using a portable sleep monitor for home use; results will be analyzed by a sleep medicine specialist. Finally, each subject will undergo a battery of performance -based cognitive function tests that measure visual and auditory memory, processing speed, attention, and eye-hand coordination. If magnetic resonance imaging (MRI) evaluation has been performed within the past 5 years, the film will be reviewed by a neuroradiologist to assess the presence of white matter lesions. Additional MRI will not be performed as part of the study. Completion of the study will necessitate up to three clinic visits (total 5-6 hours) and the home sleep study.

The research questions are as follows:

* Does the presence of a large PFO have any impact on cognitive function, particularly in brain regions supplied by posterior circulation, in migraine aura?
* Does cerebral vasomotor reactivity differ between migraineurs with aura, with and without large PFO?
* Do migraineurs with aura and large PFO have higher biomarkers of platelet activation (soluble P-selectin, sCD40L, TXB2) than migraineurs with aura without PFO?
* Are there differences in the prevalence and severity of sleep apnea, as assessed by apnea-hypopnea index (AHI), in migraine aura, with and without large PFO?
* What is the effect of large PFO on monthly migraine frequency (MMF) and aura frequency?

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years
2. Ability to speak, read, and understand English
3. Documented diagnosis of migraine aura (MA) for a ≥2 year period preceding enrollment, confirmed by a neurology healthcare provider (MD, DO, ARNP, PA-C) using the International Classification of Headache Disorders criteria. Focal neurologic symptoms must precede or accompany the headache (aura) for at least one headache in the 12 months prior to enrollment.
4. Average of 4 to 14 migraine days per month for the 3-month period preceding enrollment
5. Migraine prevention regimen stable for at least 30 days prior to enrollment. This criterion does not pertain to acute medications or aspirin- or non-steroidal anti-inflammatory (NSAID)- containing medications, which will be held (wash-out) prior to blood draw. See below.
6. Able and willing to complete a washout of aspirin, NSAIDs (including ibuprofen, naproxen sodium, ketorolac), combination drugs containing these compounds, or dietary supplements containing willow bark (salicylate) prior to blood collection.
7. Experimental group: Documented large right-to-left shunt (RLS) with >100 embolic tracks (ET) at rest or following calibrated or uncalibrated respiratory strain by TCD (whichever yields largest number of ET).
8. Control group: Documented absence of right-to-left shunt (RLS) with <11 ET at rest and following calibrated and uncalibrated respiratory strain by TCD (whichever yields largest number of ET).
9. Adequate correction of hearing and/or vision deficits

Exclusion Criteria:

1. Pregnancy
2. Postmenopausal female
3. Documented right-to-left shunt (RLS) with 11 to 100 ET at rest or following calibrated or uncalibrated respiratory strain by TCD (whichever yields largest number of ET)
4. History of stroke or neurological condition associated with cognitive dysfunction such as multiple sclerosis, epilepsy, brain tumor or brain injury
5. Chronic migraine or medication overuse headache
6. Prescription use of warfarin or antiplatelet drug such as clopidogrel or aspirin
7. Inability or unwillingness to complete a washout of aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), combination drugs containing these compounds, or dietary supplements containing willow bark (salicylate)
8. Evidence of carotid, vertebral, or basilar artery stenosis >50% on duplex imaging
9. Evidence of fetal origins or >50% stenosis of intracranial blood vessels on TCD imaging
10. Inadequate temporal bone windows (signals) for TCD insonation
11. Daily treatment regimen includes topiramate and/or other medication that causes significant cognitive or psychomotor impairment based on provider assessment and/or self-report (e.g., amitryptiline, divalproex sodium)
12. Use of continuous positive-airway pressure (CPAP) instrumentation within 6 months of study enrollment
13. Status post PFO or RLS closure/repair
14. Beck Depression Inventory score ≥29
15. State-Trait Anxiety Inventory score exceeding cutoff for age and sex

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Otherwise healthy persons who have a diagnosis of MA, based on the International Classification of Headache Disorders Diagnostic Criteria, will be recruited from headache and neurology clinics. Potential subjects can self refer if they have a diagnosis of MA.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill T. Jesurum, Ph.D., Principal Investigator — Swedish Medical Center; Cindy J. Fuller, Ph.D., Principal Investigator — Swedish Medical Center; Sylvia M. Lucas, M.D., Ph.D., Study Chair — University of Washington; Natalia Murinova, M.D., Study Chair — University of Washington; Alan M. Haltiner, Ph.D., Study Chair — Swedish Medical Center; Colleen M. Douville, B.S., Study Chair — Swedish Medical Center
Locations (2):
- United States (2):
  - Swedish Medical Center, Seattle, Washington
  - The University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over a 20-month period (January 2010 to May 2011), 127 subjects were screened and 31 were enrolled from Swedish Medical Center and the University of Washington Medical Center, including 19 with MA + PFO and 12 with MA - PFO.
Pre-assignment Details: Of 127 potential subjects screened, reasons for exclusion included the following:
  22 (17%) chronic migraine or medication overuse headache; 9 (7%) topiramate use; 6 (5%) stroke or multiple sclerosis; 39 (31%) other (declined, low frequency); 12 (9%) small to medium sized PFO; 8 (6%) fetal origins.
Period: Overall Study
Arm/Group | Control (Absence of PFO) | Large PFO
Started | 12 | 19
Completed | 12 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Absence of PFO) | Large PFO | Total
Number analyzed (Participants) | 12 | 19 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 19 | 31
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (10) | 35 (11) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Embolic Tracks
Description: Embolic tracks on transcranial Doppler at rest and following calibrated Valsalva maneuver
Time Frame: Baseline
Reporting Status: Not Posted

2. Primary Outcome: Cerebral Vasomotor Reactivity (VMR)
Description: The percentage change in basilar artery blood flow velocity from baseline between hypercapnia (increased blood CO2) and hypocapnia (decreased blood CO2), as measured by transcranial Doppler during a single testing period. This is calculated using the following equation:
  VMR = 100 x (VelocityHYPERCAPNIA - VelocityHYPOCAPNIA) / VelocityBASELINE
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Control (Absence of PFO) | Large PFO
Number analyzed (Participants) | 12 | 19
Percentage change | 89 (20) | 97 (24)
Statistical Analysis 1: Comparison: Control (Absence of PFO) vs Large PFO; Mann-Whitney U test was used to test the null hypothesis that basilar artery vasomotor reactivity was equivalent between the two groups; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Platelet Activation
Description: Platelet-poor plasma levels of sCD40L and P-selectin, and serum concentration of TXB2.
Time Frame: Baseline
Reporting Status: Not Posted

4. Primary Outcome: Sleep Apnea, Number of Participants
Description: An apnea-hypopnea index (AHI) >10 per hour during a home sleep study, defined as at least 5 hours of recorded data on the portable sleep monitor instrument for either the apnea-hypopnea index (AHI) or oxygen desaturation index (ODI) and at least 3 hours for the other index. The scale adopted for assessment of sleep apnea is as follows: AHI < 5, optimal; AHI 5-10, equivocal, participant may have sleep apnea; AHI >10, sleep apnea highly likely.
Time Frame: Following one night of a home sleep study
Population: The analysis was based on per protocol.
Measure: Number; unit: participants
Arm/Group | Control (Absence of PFO) | Large PFO
Number analyzed (Participants) | 11 | 16
participants | 0 | 1

5. Primary Outcome: Cognitive Function
Description: Cognitive function will be assessed by a battery of performance-based neuropsychological tests.
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Oxygen Desaturation Index
Description: Measurement of number of times per hour blood oxygen saturation decreases by at least 4% during home sleep study.
Time Frame: Baseline
Reporting Status: Not Posted

7. Secondary Outcome: White Matter Lesions
Description: Presence and severity of white matter lesions on magnetic resonance imaging, taken within 5 years prior to study enrollment. Subjects will not have magnetic resonance imaging performed as part of this study. Films will be requested and an independent neuroradiologist will assess presence of white matter lesions.
Time Frame: Within 5 years prior to enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control (Absence of PFO) | Large PFO
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/19
Other Adverse Events (participants affected / at risk) | 0/12 | 0/19

LIMITATIONS AND CAVEATS:
Subjects were recruited from a headache clinic and had a high degree of migraine burden; thus, the sample may not accurately represent the general migraine population. The number of men in the sample was insufficient to test sex differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No